CLINICAL TRIAL: NCT06888635
Title: Predicting the Metabolic Biomarkers Associated With Injury in Athletes
Status: Enrolling by invitation | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-25-003
Record Dates: First submitted 2025-03-02; First posted 2025-03-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-03

CONDITIONS: Sports Medicine
Keywords: sports medicine,; injury; biomarker; metabolite
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute Injury athletes: Athletes in sports, due to sudden external force or improper operation, resulting in body tissue damage in a short period of time. This injury usually has sudden and distinct traumatic features, and common types include:
  1. Sprain: Joint due to excessive torsion or stretching, resulting in ligament damage.
  2. Strain: An injury to a muscle or tendon caused by excessive stretching or contraction.
  3. Contusion: A direct impact on the body part causes damage to the subcutaneous tissue, which may be accompanied by bruising.
  4. Fracture: The bone is broken due to external force.
  5. Dislocation: The joint is removed from its normal position due to external forces.
- Healthy athletes: athletes with no acute injury in the last 3 months
- Healthy: Healthy non-athlete population

SUMMARY:
For elite athletes, sports injuries significantly impede the further enhancement of their competitive performance. Consequently, the significance of preventing, detecting, and addressing potential injury issues has become increasingly critical. Currently, the comprehensive evaluation of athletes' physical function and condition primarily depends on a range of physiological, biochemical, and immunological indicators. However, these methods have progressively exposed their limitations. As an advanced bioinformatics technology, omics research demonstrates unique advantages. By leveraging multi-omics research and analysis, it is possible to more accurately observe the physiological and biochemical changes that athletes undergo during training and competition, as well as their regulatory mechanisms. This approach can provide practical data, identify biomarkers that can warn of potential injuries, and offer precise guidance for training monitoring and injury prevention. It also provides a foundation for developing diverse, precise, and personalized sports programs and rehabilitation plans.

DETAILED DESCRIPTION:
Investigators will collect fasting venous blood. White blood cell count, red blood cell count, erythrocyte specific volume, hemoglobin, C-reactive protein, procalcitonin, erythrocyte sediment rate, lactic acid,creatine kinase, liver function indicators, blood urea, blood creatinine, blood uric acid, blood testosterone, blood cortisol, immunoglobulin (IgG, IgA, IgM) and ferritin levels were measured. The levels of IL-2, IL-6, IL-1β and TNF-α were determined by ELISA. Blood samples were purified and analyzed by proteomics, metabolomics and lipidomics methods. Urine and stool samples were collected and analyzed by multi-omics method.

ELIGIBILITY:
Inclusion Criteria:

1. Age： Athletes 12-30 years old
2. Acute injury during exercise: such as muscle, sprain, contusion, torn ligament, dislocation, fracture.

Exclusion Criteria:

1. Athletes with serious cardio-cerebrovascular disease and abnormal liver and kidney function
2. Recent use of drugs or supplements that affect metabolism.
3. Pregnancy, lactation or special conditions that may affect metabolism.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Athletes in sports, due to sudden external force or improper operation, resulting in body tissue damage in a short period of time. This injury usually has sudden and distinct traumatic features, and common types include:
  1. Sprain: Joint due to excessive torsion or stretching, resulting in ligament damage.
  2. Strain: An injury to a muscle or tendon caused by excessive stretching or contraction.
  3. Contusion: A direct impact on the body part causes damage to the subcutaneous tissue, which may be accompanied by bruising.
  4. Fracture: The bone is broken due to external force.
  5. Dislocation: The joint is removed from its normal position due to external forces.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with athletes with acute injuries | 1year
  Acute injuries are defined as the injuries of body tissues in a short period of time due to sudden external force or improper operation during sports.This injury usually has sudden and distinct traumatic features

CONTACTS AND LOCATIONS:
Overall Officials: Yue Zhang, Doctor, Principal Investigator — Department of Respiratory, Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of Respiratory, Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine,China, Shanghai, China